CLINICAL TRIAL: NCT00193154
Title: A Phase II Trial of Tarceva (OSI-774) and Avastin (Bevacizumab) in the Treatment of Patients With Metastatic Renal Cell Carcinoma
Brief Title: OSI-774 and Bevacizumab in the Treatment of Patients With Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: AstraZeneca (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GU 17; AVF2488s
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Kidney Cancer
Keywords: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Erlotinib Hydrochloride; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OSI-774 & bevacizumab (Experimental): OSI-774 (Tarceva) 150mb PO, days 1-28; bevacizumab (Avastin) 10mg/kg, IV infusion, days 1 and 15; Regimen will be repeated every 28 days.
  Interventions: Drug: OSI-774; Drug: Bevacizumab

INTERVENTIONS:
Drug: OSI-774 — 150mg PO, days 1-28, cycle repeated every 28 days
  Other Names: Tarceva
Drug: Bevacizumab — 10mg/kg, IV infusion, Days 1 and 15, 28 day cycles
  Other Names: Avastin

SUMMARY:
In this phase II trial, we plan to evaluate the combination of Tarceva and Avastin in the treatment of patients with metastatic renal cell carcinoma. This trial will be one of the first phase II trials to evaluate a combination of targeted agents in the treatment of a common solid tumor with a strong biologic rationale based on Cancer Biology (VHL/HIF/VEGF/EGFr).

DETAILED DESCRIPTION:
Upon determination of eligibility, all patients will receive:

Tarceva + Avastin

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Metastatic or unresectable clear cell kidney cancer confirmed by biopsy
* Previous nephrectomy
* Maximum of 1 previous regimen for metastatic disease
* Ability to perform activities of daily living with minimal assistance
* Measurable disease
* Adequate bone marrow, liver and kidney function
* Give written informed consent prior to study entry

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Age < 18 years
* Treatment with more than one previous regimen for metastatic disease
* Clinically significant cardiovascular disease
* Active brain metastases
* History of CNS disease
* Clinical history of coughing or vomiting blood.
* History of thromboembolic disease.
* PEG or G-tube are ineligible.
* Current use of full dose anticoagulants or thrombolytic agents
* Chronic daily treatment with aspirin or NSAIDS
* Any clinical evidence or history of a bleeding or clotting disorder

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2003-02; Primary Completion 2004-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of the combination of Tarceva and Avastin | 18 months

SECONDARY OUTCOMES:
Objective response rate | 18 months
Progression-free survival | 18 months
Overall Survival | 18 months
Overall tolerability and toxicity of this combination regimen | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (2):
- United States (2):
  - Medical Oncology LLC, Baton Rouge, Louisiana
  - Grand Rapids Oncology Program, Grand Rapids, Michigan

REFERENCES:
- [Result] Hainsworth JD, Sosman JA, Spigel DR, Edwards DL, Baughman C, Greco A. Treatment of metastatic renal cell carcinoma with a combination of bevacizumab and erlotinib. J Clin Oncol. 2005 Nov 1;23(31):7889-96. doi: 10.1200/JCO.2005.01.8234. Epub 2005 Oct 3. PMID 16204015
- See also: Published article in the Journal of Clinical Oncology — http://jco.ascopubs.org/cgi/reprint/23/31/7889